CLINICAL TRIAL: NCT07249047
Title: Correlation Between Optic Nerve Sheath Diameter Measured by Ultrasound and Delirium in Cardiac Surgery
Brief Title: Association of Optic Nerve Sheath Diameter and Postoperative Delirium
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Mauricio Giraldo, Anesthesiologist, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONSD & Delirium
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Delirium
Keywords: Post operative delirium; Optic nerve sheath diameter; Anesthesia
MeSH Terms: conditions — Emergence Delirium | interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Optic nerve sheath diameter (ONSD) ultrasound
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optic nerve sheath diameter (ONSD) ultrasound (Experimental): Optic nerve sheath diameter (ONSD) ultrasound to be performed at the following time points:
  1. Prior to the start of surgery
  2. At the start of cardiopulmonary bypass (CPB)
  3. At the end of cardiopulmonary bypass
  4. Admission to the ICU
  5. 1 hour after ICU admission
  6. 6 hours after ICU admission
  7. 24 hours after ICU admission
  8. Daily until hospital discharge for delirious patients or daily until discharge from the ICU for non-delirious patients.
  Delirium will be assessed by administering the Intensive Care Delirium Screening Checklist (ICDSC) to patients twice daily until discharge from ICU.
  Interventions: Procedure: Optic nerve sheath diameter (ONSD) ultrasound

INTERVENTIONS:
Procedure: Optic nerve sheath diameter (ONSD) ultrasound — Optic nerve sheath diameter (ONSD) ultrasound to be performed to measure diameter of the optic nerve sheath. Administration of the Intensive Care Delirium Screening Checklist (ICDSC) twice daily until discharge from the ICU.

SUMMARY:
Postoperative delirium is a sudden and reversible disturbance of mental function, occurring after surgery, characterized by confusion, inattention, and fluctuating mental status, which can manifest as agitation or lethargy. It is a common post-operative complication, especially in older adults, and is associated with longer hospital stays and worse recovery outcomes. Validated delirium screening tools such as the Intensive Care Delirium Screening Checklist (ICDSC) and the Richmond Agitation and Sedation Scale (RASS) are widely used tools to assess delirium. However, the sensitivity of these screening tools can be variable when used in real-world practice and may miss early cases of delirium. The optic nerve sheath is a protective sheath that encloses part of the optic nerve that is located at the back of the eye. Measurement of the optic nerve sheath diameter is usually done using ultrasound to detect increased cranial pressure. Previous studies that have been conducted have shown that increased ONSD may be associated with occurrence of postoperative delirium. The purpose of this study is to determine if there is an association between optic nerve sheath diameter (ONSD) and the occurrence of delirium after surgery. This study will be conducted at the London Health Sciences Centre and will include 300 patients.

DETAILED DESCRIPTION:
Delirium is one of the most frequent and serious complications after cardiac surgery, with reported incidence between 15-30% depending on patient population, procedure type, and diagnostic method. It is associated with prolonged ICU and hospital length of stay, increased risk of institutional discharge, higher readmission rates, long-term cognitive impairment, and mortality. Validated delirium screening tools such as the Confusion Assessment Method for the ICU (CAM-ICU) and the Intensive Care Delirium Screening Checklist (ICDSC) are widely used, but their sensitivity in real-world practice can be variable, sometimes missing early cases despite high specificity. This contributes to delayed recognition and potentially worse outcomes.

Ultrasound measurement of the optic nerve sheath diameter (ONSD) has emerged as a non-invasive surrogate marker for intracranial pressure (ICP). Several meta-analyses confirm good diagnostic accuracy of ONSD ultrasound compared to invasive ICP monitoring. Concordance studies also demonstrate strong agreement between ultrasound and MRI ONSD measurements, particularly when standardized measurement protocols are used (e.g., 3 mm posterior to the retina, bilateral averaging). These findings support the reliability of ONSD ultrasound as a bedside monitoring tool.

In critical care, early broadening of ONSD has been associated with delirium, coma, and death within 28 days. Importantly, the first cardiac surgery-specific study that prospectively examined patients undergoing open-heart surgery and found that increased peri-operative ONSD was independently associated with postoperative delirium. Their findings suggest that ONSD may serve not only as a marker of raised ICP but also as a predictive biomarker for delirium in the cardiac surgical population. Taken together, the burden of postoperative delirium in cardiac surgery, the limitations of current screening methods, and the growing evidence supporting ONSD as a surrogate of cerebral dynamics provide the rationale for this study. We hypothesize that perioperative or early ICU ONSD enlargement will be associated with the development of delirium, and that ONSD monitoring may help identify high-risk patients earlier, guiding preventive strategies.

Informed, written consent will be obtained prior to the start of surgery. The participant's surgical plan will not be altered in any way. Participants that are enrolled in this study will have their surgery proceed according to plan and will be placed under general anesthesia using standard of care practices. Cardiopulmonary bypass will be implemented in accordance with standard of care practices.

For the ONSD ultrasound, the ultrasound will be performed using a linear probe 7.5-13 MHz and will follow standard practice for this procedure. Patients will have closed eyelids covered with a Tegaderm adhesive for eye protection. Ultrasound gel will be applied to the patient's eyelids. The ultrasound probe will be gently placed on the patient's eyelids and to locate the optic nerve and measure ONSD. The ultrasound scan will be performed 3 mm posterior to retina with 4 measurements taken at each time point to allow for a mean result to be determined. Average time for each measurement is 1 minute. Each ultrasound will take 10-15 minutes to complete. This ONSD ultrasound will be performed at the following time points:

1. Prior to the start of surgery
2. At the start of cardiopulmonary bypass (CPB)
3. At the end of cardiopulmonary bypass
4. Admission to the ICU
5. 1 hour after ICU admission
6. 6 hours after ICU admission
7. 24 hours after ICU admission
8. Daily until hospital discharge for delirious patients or daily until discharge from the ICU for non-delirious patients.

Delirium will be assessed by administering the Intensive Care Delirium Screening Checklist (ICDSC) to patients twice daily until discharge from ICU. This ICDSC will be administered in person. The study team will also collect information such as the patient's age, biological sex, height, weight, medications, medical history, surgical details, results of preoperative and postoperative blood work, pain scores that are collected as part of standard of care practices, and details of their postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* A d u l t s ≥ 1 8 y e a r s .
* Scheduled for cardiac surgery requiring cardiopulmonary bypass (CPB) (e.g., Coronary artery bypass graft (CABG), valve, combined procedures, aortic surgery).
* Anticipated postoperative admission to the Cardiac ICU with expected stay >48 hours.
* Preoperative ability to undergo ocular ultrasound examination (closed-eyelid scanning).
* Provided informed consent to participate in this study.

Exclusion Criteria:

* Known or suspected open-globe injury, penetrating ocular trauma, or intraocular foreign body.
* Recent ocular surgery or intravitreal intervention within the past 6 weeks (if surgeon advises against periocular pressure).
* Ocular conditions that invalidate ONSD measurement (e.g., severe proptosis, advanced optic neuropathies, orbital tumors) or obstruct ultrasound window (extensive periocular dressings, severe periorbital edema).
* Known intracranial pathology expected to significantly alter baseline ONSD (e.g., large mass lesion with midline shift, obstructive hydrocephalus) or presence of external ventricular drain at baseline.
* Severe facial trauma or unstable cervical spine precluding safe positioning for ocular ultrasound.
* P r e g n a n c y .
* Inability to perform serial ONSD assessments at scheduled timepoints (e.g., continuous prone positioning) despite reasonable accommodations.
* Enrollment in a conflicting interventional trial that mandates deviations from delirium assessment or ONSD protocol.
* Inability to communicate in the English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of optic nerve sheath diameter on postoperative delirium | Days 1-3 postoperatively
  This will be measured by comparing the diameter of the optic nerve sheath to the results of the Intensive Care Delirium Screening Checklist (ICDSC) that will be used to measure delirium in patients. The ICDSC will provide a score of 0-8 for patients. Scores of 4 or higher will be considered to be indicative of postoperative delirium.

SECONDARY OUTCOMES:
Impact of optic nerve sheath diameter on hospital length of stay | Days 1-7 postoperatively
  This will be measured by noting how long the patient is in hospital following surgery and comparing that to optic nerve sheath diameter.
Impact of optic nerve sheath diameter on mortality | Days 1-7 postoperatively
  This will be measured by noting if a participant has died and comparing that to optic nerve sheath diameter.
Impact of optic nerve sheath diameter on time spent on a ventilator | Days 1-7 postoperatively
  This will be measured by noting how long the patient is required to use a ventilator (if applicable) following surgery and comparing that to optic nerve sheath diameter.
Impact of optic nerve sheath diameter on the need for re-intubation | Days 1-7 postoperatively
  This will be measured by noting if a participant requires re-intubation following surgery and comparing that to optic nerve sheath diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Giraldo, MD, Principal Investigator — London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mattimore D, Fischl A, Christophides A, Cuenca J, Davidson S, Jin Z, Bergese S. Delirium after Cardiac Surgery-A Narrative Review. Brain Sci. 2023 Dec 7;13(12):1682. doi: 10.3390/brainsci13121682. PMID 38137130
- [Background] Koster S, Hensens AG, Schuurmans MJ, van der Palen J. Consequences of delirium after cardiac operations. Ann Thorac Surg. 2012 Mar;93(3):705-11. doi: 10.1016/j.athoracsur.2011.07.006. Epub 2011 Oct 10. PMID 21992939
- [Background] Mangusan RF, Hooper V, Denslow SA, Travis L. Outcomes associated with postoperative delirium after cardiac surgery. Am J Crit Care. 2015 Mar;24(2):156-63. doi: 10.4037/ajcc2015137. PMID 25727276
- [Background] Chen H, Mo L, Hu H, Ou Y, Luo J. Risk factors of postoperative delirium after cardiac surgery: a meta-analysis. J Cardiothorac Surg. 2021 Apr 26;16(1):113. doi: 10.1186/s13019-021-01496-w. PMID 33902644
- [Background] van Eijk MM, van den Boogaard M, van Marum RJ, Benner P, Eikelenboom P, Honing ML, van der Hoven B, Horn J, Izaks GJ, Kalf A, Karakus A, Klijn IA, Kuiper MA, de Leeuw FE, de Man T, van der Mast RC, Osse RJ, de Rooij SE, Spronk PE, van der Voort PH, van Gool WA, Slooter AJ. Routine use of the confusion assessment method for the intensive care unit: a multicenter study. Am J Respir Crit Care Med. 2011 Aug 1;184(3):340-4. doi: 10.1164/rccm.201101-0065OC. Epub 2011 May 11. PMID 21562131
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Robba C, Santori G, Czosnyka M, Corradi F, Bragazzi N, Padayachy L, Taccone FS, Citerio G. Optic nerve sheath diameter measured sonographically as non-invasive estimator of intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2018 Aug;44(8):1284-1294. doi: 10.1007/s00134-018-5305-7. Epub 2018 Jul 17. PMID 30019201
- [Background] Dubourg J, Javouhey E, Geeraerts T, Messerer M, Kassai B. Ultrasonography of optic nerve sheath diameter for detection of raised intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2011 Jul;37(7):1059-68. doi: 10.1007/s00134-011-2224-2. Epub 2011 Apr 20. PMID 21505900
- [Background] Shirodkar CG, Munta K, Rao SM, Mahesh MU. Correlation of measurement of optic nerve sheath diameter using ultrasound with magnetic resonance imaging. Indian J Crit Care Med. 2015 Aug;19(8):466-70. doi: 10.4103/0972-5229.162465. PMID 26321806
- [Background] Steinborn M, Fiegler J, Ruedisser K, Hapfelmeier A, Denne C, Macdonald E, Hahn H. Measurement of the Optic Nerve Sheath Diameter in Children: Comparison Between Transbulbar Sonography and Magnetic Resonance Imaging. Ultraschall Med. 2012 Dec;33(6):569-573. doi: 10.1055/s-0031-1273491. Epub 2011 Aug 25. PMID 21870318
- [Background] Zhi H, Cui X, Zhang F, Wang S, Liang X, Wang B, Cui J, Li Y. [Bedside ultrasound monitoring of optic nerve sheath diameter is a predictive factor for 28-day coma, delirium and death in etiologically diverse critically ill patients]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2024 Oct;36(10):1088-1094. doi: 10.3760/cma.j.cn121430-20230511-00362. Chinese. PMID 39586729
- [Background] Kaynar A, Komurcu O, Bahsi E, Aydin AO, Karal IH, Akyurt D, Tulgar S, Suren M. Optic nerve sheath diameter is associated with postoperative delirium in patients undergoing open heart surgery. BMC Anesthesiol. 2025 Jul 1;25(1):309. doi: 10.1186/s12871-025-03194-9. PMID 40596877
- [Background] Mount CA, Das JM. Cerebral Perfusion Pressure. 2023 Apr 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537271/ PMID 30725956
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Background] Vittinghoff E, McCulloch CE. Relaxing the rule of ten events per variable in logistic and Cox regression. Am J Epidemiol. 2007 Mar 15;165(6):710-8. doi: 10.1093/aje/kwk052. Epub 2006 Dec 20. PMID 17182981
- [Background] Yang H, Zhang L, Huang P, Luo Y. [Investigation of intracranial pressure in intensive care unit patients with delirium assessed by bedside ultrasound]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2022 Jun;34(6):635-639. doi: 10.3760/cma.j.cn121430-20220523-00504. Chinese. PMID 35924521
- [Background] Mowafy SMS, Bauiomy H, Kohaf NA, Abd Ellatif SE. The Role of Ultrasonographic Assessment of Optic Nerve Sheath Diameter in Prediction of Sepsis-Associated Encephalopathy: Prospective Observational Study. Neurocrit Care. 2025 Aug;43(1):308-317. doi: 10.1007/s12028-024-02187-9. Epub 2025 Jan 15. PMID 39815108